CLINICAL TRIAL: NCT04620837
Title: A Prospective, Open Label, Single-arm, Phase 2 Study of Tislelizumab in Combination With Anlotinib as Maintenance Therapy in Subject With Extensive Stage Small Cell Lung Cancer （ES-SCLC） as Maintenance Therapy After First Line Chemotherapy
Brief Title: Tislelizumab in Combination With Anlotinib With ES-SCLC as Maintenance Therapy After First Line Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-04254
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-10

CONDITIONS: Small Cell Lung Carcinoma
Keywords: Human anti-human PD-1 monoclonal antibody; Receptor Tyrosine Kinase inhibitor(RTKi)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Tislelizumab：200mg Q3W IV Anlotinib hydrochloride capsules: Capsule; specifications 12mg; oral, once a day, every 12mg, continuous medication two weeks after 1 week deactivated.
  Interventions: Drug: Tislelizumab; Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab：200mg Q3W IV. There will be no dose reduction for Tislelizumab ， if there is no disease progression or serious Treatment Related adverse events(TRAE) , patients will receive Tislelizumab (200mg,Q3W) until progression or death
Drug: Anlotinib hydrochloride — Anlotinib hydrochloride capsules: Capsule; specifications 12mg; oral, once a day, every 12mg, continuous medication two weeks after 1 week deactivated. Depending tolerated dose reduction. Medication process: disease control and patients can tolerate the side effects, continued drug use; researchers believe the patient is not fit to continue medication or efficacy evaluation at the end of the clinical progression of medication.
  Other Names: Anlotinib

SUMMARY:
To show that maintenance therapy with Tislelizumab plus Anlotinib will prolong Progression Free Survival in subjects with extensive stage disease small cell lung cancer who have completed first line chemotherapy.

DETAILED DESCRIPTION:
Most patients with extensive disease small cell lung cancer (ED-SCLC) respond to first line（1L） platinum-based chemotherapy; however, responses are not durable and prognosis is poor. Currently no maintenance treatments are approved in SCLC to prolong the durability of efficacy achieved with 1L chemotherapy. Immuno-oncology agents have demonstrated efficacy in the treatment of ED-SCLC when administered across different lines of therapy. Tislelizumab (Anti-PD-1 antibody) Combine Etoposide+ platinum （EP） had improved median Overall survival （mOS ） to 15.6m of 1L ED-SCLC in the Rationale 206 study. Anlotinib ( RTKi ) had significantly improved PFS & OS of 3L(third line) ED-SCLC in the ALTER 1202. This phase II study is designed to explore the effect and safety of the combination as maintenance therapy for ED-SCLC after 1L chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically confirmed extensive stage disease SCLC
* Ongoing response of stable disease or better following 4 cycles of platinum-based first line chemotherapy
* Patients should enter the study within 5 weeks after the completion of cycle 4 chemotherapy (the last dose).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 Extensive-stage disease at diagnosis
* Patients must have received 4 cycles of platinum-containing chemotherapy and must be at the level of complete remission (CR), partial remission (PR), or disease stabilization (SD) at the time of completion of chemotherapy. According to the The National Comprehensive Cancer Network （NCCN） guidelines, acceptable combination therapy includes cisplatin or carboplatin plus etoposide or irinotecan.
* The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 6 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 6 months after it
* Otherwise healthy

Exclusion Criteria:

* Subjects with symptomatic Central Nervous System (CNS) metastases
* Subjects receiving consolidative chest radiation
* Subjects with active, known, or suspected autoimmune disease are excluded Cancerous meningitis.
* Pleural effusions that are not controlled by appropriate interventions
* All side effects attributed to prior anti-cancer therapy must have resolved to Grade 1 or baseline
* Medical history and concurrent diseases. a) Pregnant or lactating women. b) Active, known or suspected autoimmune diseases. Exclude conditions that require immunosuppressive therapy. d) Previous use of anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibodies (including Ipilimumab or any other T-cell co-stimulation or checkpoint pathway points) The antibody or drug e). The subject has interstitial lung disease, the disease has symptoms, or the disease may affect the discovery or management of suspected drug-related lung toxicity. f) Previous malignancy unless at least prior to participating in the study Completely relieved 2 years ago and requires no additional treatment during the study. g)Based on the investigator's judgment, known medical conditions increase the risk associated with participating in the study or giving the blinded study drug or affecting the interpretation of the findings.
* Physical examination and laboratory tests found. a)Hepatitis B virus （HBV） surface antigen test to determine hepatitis B virus positive, or Hepatitis C virus（ HCV） ribonuclease test to determine hepatitis C virus positive, or HCV antibody test showed acute or chronic infection. b) A history of HIV-positive disease is known or a history of AIDS disease is known. c) Insufficient hematopoietic function. d)Insufficient liver function. e) insufficient pancreatic function
* Patients get any severe diseases or the ones that cannot be controlled take major surgical treatments, open biopsy, or get overt traumatic injury within 28 days before grouping
* Patients have any habitus or medical history of hemorrhage, however severe it is; the patients who have non healing wounds, ulcer or fracture after any events with hemorrhage or bleeding (> or =CTCAE level 3)
* Patients get arterial/venous thrombosis within 6 months, such as cerebrovascular accidents (including temporary ischemic stroke), deep venous thrombosis, and pulmonary embolism
* Patients ever abuse psychiatric drugs and cannot abstain or who are diagnosed with mental disorder
* -Patients have participated in other clinical trials of anti-tumor medicine within 4 weeks
* Patients diagnosed with disease which will severely endanger the security of patients or influence the completion of this research.
* Allergies and Adverse Drug Reactions: A history of allergies or hypersensitivity reactions to any study drug or other study drug component

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of progression free survival | 6 months
  Rate of progression free survival in 6 month

SECONDARY OUTCOMES:
overall survival | 24 months
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- National Cancer Center/Cancer Hospitial,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No